CLINICAL TRIAL: NCT06346288
Title: A Phase 4, Open-Label, Milk-Only Lactation Study to Assess Concentration of Risankizumab in Breast Milk of Lactating Women With Inflammatory Bowel Disease Who Are Receiving Risankizumab Therapeutically
Brief Title: A Study to Assess the Concentrations of Risankizumab in the Breast Milk of Adult Lactating Women With Inflammatory Bowel Disease
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M24-144
Record Dates: First submitted 2024-03-22; First posted 2024-04-04 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD; Lactating; breastfeeding; risankizumab; Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; SKYRIZI
MeSH Terms: conditions — Inflammatory Bowel Diseases; Breast Feeding; Crohn Disease; Colitis, Ulcerative | interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pharmacokinetic samples (Experimental): Pharmacokinetic (PK) samples will be taken from breast milk of lactating mothers on an established dosing regimen of commercial risankizumab at pre-dose and 1 hour after dosing on Day 1, on Days 4 (± 1), 8 (± 2), 15 (± 3), 29 (± 3), and pre-dose on Day 57 (± 3).
  Participants will have already been taking commercial risankizumab and will continue on commercial risankizumab. Participants will not be provided risankizumab from the study. Participants must have received at least 2 doses of 360 mg of risankizumab SC every 8 weeks postpartum prior to start of participation in this study.
  Interventions: Procedure: Breast Milk Sampling; Drug: Risankizumab

INTERVENTIONS:
Procedure: Breast Milk Sampling — Pharmacokinetic (PK) samples will be taken from breast milk of lactating mothers on an established dosing regimen of commercial risankizumab at pre-dose and 1 hour after dosing on Day 1, on Days 4 (± 1), 8 (± 2), 15 (± 3), 29 (± 3), and pre-dose on Day 57 (± 3)
Drug: Risankizumab — Participants will have already been taking commercial risankizumab and will continue on commercial risankizumab. Participants will not be provided risankizumab from the study. Participants must have received at least 2 doses of 360 mg of risankizumab SC every 8 weeks postpartum prior to start of participation in this study.
  Other Names: SKYRIZI

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic inflammatory disease that requires lifelong treatment. This study will asses the concentrations of risankizumab in the breast milk of lactating women with IBD

Risankizumab is an approved drug for adults with plaque psoriasis, psoriatic arthritis, and Crohn's Disease. This is an open-label milk-only study lactation study to evaluate the presence of risankizumab in the milk of lactating women. Approximately 10 adult lactating women with IBD will be enrolled from approximately 3 sites in Israel and or the United States.

Participants will receive risakizumab maintenance therapy every 8 weeks postpartum prior to start of participation in this study. The study duration is approximately 7 months.

Participants will attend regular visits during the study at a hospital or clinic. The participants will also be completing questionnaires and will have medical assessments, checking for side effects.

DETAILED DESCRIPTION:
The study will only include lactating women who are receiving treatment with risankizumab for IBD in accordance with their treating physician, although this study is non-interventional regarding treatment with risankizumab, it is considered interventional due to the collection of breast milk from the lactating mothers.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have received at least 2 doses of 360 mg risankizumab maintenance therapy every 8 weeks postpartum prior to start of participation in this study.
* Participant is at least 5 weeks postpartum by Day 1.
* Lactation is well established. The mother must be exclusively breastfeeding her infant (or not providing more than 1 supplemental bottle of formula/day) when enrolled in the study.
* Diagnosis of crohn's disease (or ulcerative colitis upon approval of ulcerative colitis in the participants location) as established by the principal investigator

Exclusion Criteria:

* Participants who have major surgery planned during the conduct of the study (e.g., hip replacement, aneurysm removal, stomach ligation)
* Participants with the following chronic or active infections:

  -- Active HBV or HCV infection, defined as:
  * HBV: HBs Ag positive (+) test or detected sensitivity on the HBV DNA PCR qualitative test for participants who are HBc Ab positive (+) (and for HBs Ab positive [+] participants where mandated by local requirements).
  * HCV: HCV RNA detectable in any subject with HCV Ab.
* Are infected with HIV, defined as confirmed positive anti-HIV Ab test. Note: In case a screened participant has a confirmed positive HIV Ab test,.
* Active tuberculosis
* Active systemic infection/clinically important infection during the last 2 weeks prior to the Baseline Visit as assessed by the investigator
* Participants who have any of the following medical diseases or conditions:

  * Recent (within past 6 months) cerebrovascular accident or myocardial infarction;
  * History of an organ transplant which requires continued immunosuppression;
  * Active or suspected malignancy or history of any malignancy within the last 5 years except for successfully treated non-melanoma skin cancer or localized carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To determine the concentration of risankizumab in breastmilk | Pre-dose and 1 hour after dosing on Day 1, on Days 4 (± 1), 8 (± 2), 15 (± 3), 29 (± 3), and pre-dose on Day 57 (± 3)
  Breastmilk samples will be collected to evaluate the presence of risankizumab in the milk of lactating women

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (3):
- United States (2):
  - University of North Carolina at Chapel Hill /ID# 263316, Chapel Hill, North Carolina
  - UTHealth Women's Research Program - Memorial City /ID# 263939, Houston, Texas
- Shaare Zedek Medical Center /ID# 262738, Jerusalem, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-144